CLINICAL TRIAL: NCT04895813
Title: The Effect of Education and Telephone Guidance Given to the Patient Before Colonoscopy on the Patient's Anxiety Level and Bowel Preparation: A Randomized Controlled Study
Brief Title: The Effect of Education and Telephone Guidance at Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Assit. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Necmettin ErbakanU
Record Dates: First submitted 2021-05-08; First posted 2021-05-20 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Patient Education; Guidance; Colonoscopy; Nursing
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Open label posttest controlled parallel group randomized controlled study
Masking Description: NO MASKING
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: (Experimental): The patient will be given training on the day the appointment is made for colonoscopy, educational material will be given as a reminder, information will be given on the phone and the training will be reminded on the day he should start diet for colonoscopy. No different application will be made on the day and after the colonoscopy.
  Interventions: Behavioral: Education
- Group 2 (No Intervention): Routine information in the service will be made

INTERVENTIONS:
Behavioral: Education — The patient will be given pre-colonoscopy training and guidance by telephone.
  Other Names: Gudiance
  Arms: Group 1:

SUMMARY:
Colonoscopy is an endoscopic procedure for diagnosing colon diseases. Patients should be prepared 2-5 days in advance for this procedure and intestinal cleansing should be provided. This is a difficult process and does not admit mistakes. The adequacy of the patient's pre-preparation for this process increases the chances of success. For preliminary preparation, it is recommended to train the patient and reinforce the trainings by phone. Education given to the patient; It contributes positively to patient outcomes, the workload of healthcare personnel in the institution, and costs. Therefore, this study has been planned.

DETAILED DESCRIPTION:
Colonoscopy is an endoscopic procedure for the diagnosis of colon diseases. For this procedure, patients should be prepared 2-5 days in advance and intestinal cleansing should be provided. Because the adequacy of bowel cleansing provides more accurate results than colonoscopy. Pre-colonoscopy preparation process for the patient; It is very tiring and challenging for reasons such as dieting, taking too much fluid and needing to defecate constantly. After this difficult preparation period, the failure to obtain sufficient imaging from the colonoscopy necessitates going back to the beginning. But patient; If he is informed about the importance of this preparation, how it should be done, medication and fluid intake, diet, and if he is guided, the chances of success in colonoscopy will increase. For this reason, nursing education to be given to the patients before colonoscopy and the guidance of the nurse will reduce the possibility of experiencing these negativities.For this reason, this study was planned as a randomized control in order to obtain results with high evidence value. Both a printed education booklet and a digital booklet will be used and guidance will be provided by phone. As a result of this study; Before the colonoscopy procedure, a material to be used in patient education will be prepared and a printed and digital educational booklet will be provided to Necmettin Erbakan University. With the completion of the colonoscopy procedure in one go: the drugs to be used will not be prescribed repeatedly, no extra medication will be used, the patient will not be given multiple colonoscopy appointments and the procedure will not be repeated. In this way, the workload of physicians and nurses will not increase and the comfort of the patient will not be adversely affected. All of these will provide cost effective results and positive patient outcomes. Publication of the article will contribute to the literature.For this purpose, power analysis was performed, sample size was determined, and a randomization list was created for the participants. It has been planned in accordance with CONSORT. There will be 40 people in the experimental and control groups. The effect size of the study; 0.83, margin of error; 0.05 & power; It is 95%.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 18-65

* Being open to communication and cooperation
* Being conscious and in a position to answer questions
* Volunteering to research

Exclusion Criteria:

Having a disease that may affect decision making ability (dementia, psychological disorders etc.)

* Having sensory losses such as vision and hearing Colonoscopy decision has been made because of emergency and active lower gastro intestinal system bleeding.
* Being inpatient at the hospital
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The patient's anxiety level is low | Just before the colonoscopy
  It will be evaluated by the nurse before the colonoscopy procedure. State anxiety scale will be used in evaluation.The scale scores between 20 and 80, the higher the score, the higher the anxiety level
Hull cleaning of the patient's intestines and obtaining a quality image | when doing a colonoscopy
  It will be evaluated by the physician performing the procedure during the colonoscopy procedure. The image obtained from the colonoscope will be evaluated by comparing it with the bowel cleaning scale.
The patient is discharged earlier from the hospital | immediately after the colonoscopy
  It refers to the time when the patient is able to go home after the colonoscopy procedure is completed. The patient should feel completely well and there should be no problems with his vital signs. It shows how long the patient is eligible to be discharged after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Univercity, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided upon completion of the study.